CLINICAL TRIAL: NCT00775060
Title: Maastricht IBS Cohort: Phenotypical and Genotypical Characterization of Patients With Irritable Bowel Syndrome.
Brief Title: Maastricht IBS Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MEC 08-3-066
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To set up a cohort of at least 400 IBS patients in order to identify different patient subgroups according to phenotypical and genotypical patterns and

To set up a biobank for future translational studies on the pathophysiology of IBS, in order to identify genetic factors to unravel the pathogenesis of IBS and to provide novel therapeutic targets.

DETAILED DESCRIPTION:
Aim of the present study is to set up a large cohort of IBS patients in order to identify different disease characteristics as well as aetiological and pathophysiological factors in (sub)groups of patients with this heterogeneous disorder. Various phenotypical and genotypical markers will be evaluated. For this purpose, blood and faecal samples as well as symptom questionnaires will be collected and visceral perception and intestinal permeability will be measured. In order to increase the sensitivity of the barostat procedure, a pilot study will be performed by measuring patients and healthy controls under meal stimulated and fasting conditions. We aim to set up a biobank for studies on the pathophysiology of IBS, in order to identify genetic factors that may help unravel the pathogenesis of IBS and provide novel therapeutic targets. Consent will be asked to collect data from questionnaires, to store serum samples, DNA, stool and, when endoscopy is performed for clinical reasons, also biopsy specimens.

ELIGIBILITY:
Inclusion Criteria:

* IBS-patients

Exclusion Criteria:

* Severe co-morbidity hindering a rectal barostat procedure, according to the gastroenterologist's perception.
* Abdominal surgery, except for uncomplicated appendectomy, laparoscopic cholecystectomy or hysterectomy.
* Inability to stop medication that can influence gastrointestinal motility or perception (like loperamide, butylscopolamine, psylliumsead (metamucil), duspatal, metoclopramide, domperidon, erytromycin and serotonin reuptake inhibitors), for at least 3 days before tests.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 400 patients with (suspected) IBS referred to the GI-outpatient clinic of the Maastricht University Medical Center will be asked to participate in the study.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-09; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, MD, PhD, Study Director — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Snijkers JTW, Winkens B, Weerts ZZRM, Vork L, Mujagic Z, Hesselink MAM, Leue C, Kruimel JW, Muris JWM, Jonkers DMAE, Masclee AAM, Keszthelyi D. Satisfaction With Life in IBS Is Associated With Psychological Burden Rather than Gastrointestinal Symptom Severity. Am J Gastroenterol. 2024 Mar 1;119(3):512-520. doi: 10.14309/ajg.0000000000002547. Epub 2023 Oct 4. PMID 37791610
- [Derived] Vork L, Penders J, Jalanka J, Bojic S, van Kuijk SMJ, Salonen A, de Vos WM, Rajilic-Stojanovic M, Weerts ZZRM, Masclee AAM, Pozuelo M, Manichanh C, Jonkers DMAE. Does Day-to-Day Variability in Stool Consistency Link to the Fecal Microbiota Composition? Front Cell Infect Microbiol. 2021 Jul 20;11:639667. doi: 10.3389/fcimb.2021.639667. eCollection 2021. PMID 34458156
- [Derived] Mujagic Z, Jonkers DMAE, Ludidi S, Keszthelyi D, Hesselink MA, Weerts ZZRM, Kievit RN, Althof JF, Leue C, Kruimel JW, van Schooten FJ, Masclee AAM. Biomarkers for visceral hypersensitivity in patients with irritable bowel syndrome. Neurogastroenterol Motil. 2017 Dec;29(12). doi: 10.1111/nmo.13137. Epub 2017 Jul 3. PMID 28675524